CLINICAL TRIAL: NCT06823934
Title: Evaluation of the Effects of A-Prf and Oral Dexamethasone Use on Postoperative Complications in Third Molar Tooth Extraction
Brief Title: Evaluation of the Effects of A-Prf and Oral Dexamethasone Use in Third Molar Extraction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Responsible Party: Principal Investigator, Serap Keskin Tunc, Associate Professor, Yuzuncu Yil University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: YYU-13/20.09.2021
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Wisdom Tooth Removal
Keywords: Third Molar A-PRF; Dexamethasone; Postoperative Complication
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oral Dexamethasone (Active Comparator): After the extraction of the impacted wisdom tooth, the patient was prescribed oral dexamethasone (Dekort 4mg tablet, S:3*1 DEVA brand) for 3 days.
  Interventions: Procedure: Impacted lower wisdom tooth extraction
- A-Prf (Active Comparator): A-PRF was placed in the patients' tooth extraction sockets and the flap was closed primarily using 3/0 silk sutures.
  Interventions: Procedure: Impacted lower wisdom tooth extraction

INTERVENTIONS:
Procedure: Impacted lower wisdom tooth extraction — One of the most common operations performed in oral surgery is the extraction of lower impacted wisdom teeth. The extraction of impacted third molars causes significant inflammatory changes resulting in edema, trismus and pain. Complications encountered after the extraction of lower impacted wisdom teeth can negatively affect the daily lives of patients. Some of the treatments applied for these complications can be listed as drug use, cold/hot compression, low-dose laser therapy, cryotherapy, autogenous biomaterials such as PRF.

SUMMARY:
Impacted third molar tooth extraction is one of the most frequently performed procedures in oral surgery. Complications such as pain, swelling and trismus, which are frequently seen after this operation, affect the patient's quality of life in the postoperative period. Today, there are many methods used to prevent or treat these complications. Corticosteroid use and A-PRF biomaterial obtained from the patient's own blood are some of these methods. In patients with bilaterally impacted lower wisdom teeth, A-PRF was applied to one side after extraction and postoperative oral dexamethasone was used to the other side. Intra-group and inter-group evaluations were made by collecting the patients' pain, edema, trismus and analgesic use data.

DETAILED DESCRIPTION:
Impacted third molar tooth extraction is one of the most commonly performed procedures in oral surgery. Complications such as pain, swelling and trismus, which are frequently seen after this operation, affect the quality of life of the patient in the postoperative period and may cause patients to avoid this procedure. Today, there are many methods used to prevent or treat these complications. The use of corticosteroids and the A-PRF biomaterial obtained from the patient's own blood are some of these methods. No study has been found in the literature comparing the effects of oral use of dexamethasone, a corticosteroid drug, with A-PRF on pain, edema, trismus and analgesic use. In patients with bilateral impacted lower wisdom teeth, A-PRF was applied to the extraction site after extraction on one side and postoperative oral dexamethasone was used on the other side. Pain, edema, trismus and analgesic use data of the patients were collected and in-group and intergroup evaluations were made.

ELIGIBILITY:
Inclusion Criteria:

* Not having any systemic disease,
* Being over 18 years of age,
* Bilateral teeth being in similar positions and being completely impacted,
* Not having any allergies to the drugs to be used in the study.

Exclusion Criteria:

* Infection in the area where the extraction will be performed,
* Pregnancy or breastfeeding,
* Using medication up to 2 weeks before tooth extraction,
* Not using prescribed medications regularly,
* Not coming to regular check-ups.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-10-04 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-09-15 (Actual)

PRIMARY OUTCOMES:
Maximum Mouth Opening | Preoperative and postoperative 2nd, 7th, 14th and 30th days
  For the evaluation of the maximum mouth opening of the patients, the maximum mouth opening and the distance between the incisal edges of the central teeth in the most open position of the mouth were measured before the operation, on the 2nd day after the operation, on the 7th day, 14th day and 30th day after the operation.
Edema | Preoperative and postoperative 2nd, 7th, 14th and 30th days
  For the evaluation of edema of the patients, face measurements between angulus-tragus, angulus-lateral canthus, angulus-nasal wing, angulus-labial commissure, and angulus-pogonion were made before the operation, on the 2nd day after the operation, on the 7th day, 14th day, and 30th day after the operation.
VAS Pain Scor | Post-operative 3, 6, 9, 12, 24 hours and 2, 3, 4, 5, 6, 7, 14 and 30 days
  The VAS scale was used to assess the pain of the patients. Patients were instructed on how and at what time to fill out the scale, and were asked to fill out the scores from 0 to 10 (0, no pain; 10, unbearable pain) at hours 3, 6, 9, 12, and 24 and days 2, 3, 4, 5, 6, 7, 14, and 30. In order to assess the analgesic use of the patients, they were asked to note their additional analgesic use on the forms given to them.
Analgesic Consumption | Post-operative 3, 6, 9, 12, 24 hours and 2, 3, 4, 5, 6, 7, 14 and 30 days
  In order to evaluate the patients' analgesic use, patients were asked to note their additional analgesic use on the forms given to them.

CONTACTS AND LOCATIONS:
Locations (1):
- Van Yüzüncü Yıl Üniversitesi Diş Hekimliği Fakültesi, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bayer A, Wijaya B, Mobus L, Rademacher F, Rodewald M, Tohidnezhad M, Pufe T, Drucke D, Glaser R, Harder J. Platelet-Released Growth Factors and Platelet-Rich Fibrin Induce Expression of Factors Involved in Extracellular Matrix Organization in Human Keratinocytes. Int J Mol Sci. 2020 Jun 20;21(12):4404. doi: 10.3390/ijms21124404. PMID 32575800
- [Background] Pavlovic V, Ciric M, Jovanovic V, Trandafilovic M, Stojanovic P. Platelet-rich fibrin: Basics of biological actions and protocol modifications. Open Med (Wars). 2021 Mar 22;16(1):446-454. doi: 10.1515/med-2021-0259. eCollection 2021. PMID 33778163
- [Background] Selvido DI, Bhattarai BP, Niyomtham N, Riddhabhaya A, Vongsawan K, Pairuchvej V, Wongsirichat N. Review of dexamethasone administration for management of complications in postoperative third molar surgery. J Korean Assoc Oral Maxillofac Surg. 2021 Oct 31;47(5):341-350. doi: 10.5125/jkaoms.2021.47.5.341. PMID 34713808
- [Background] Moore RA, Derry S, Wiffen PJ, Straube S, Aldington DJ. Overview review: Comparative efficacy of oral ibuprofen and paracetamol (acetaminophen) across acute and chronic pain conditions. Eur J Pain. 2015 Oct;19(9):1213-23. doi: 10.1002/ejp.649. Epub 2014 Dec 22. PMID 25530283
- [Background] Bailey E, Worthington HV, van Wijk A, Yates JM, Coulthard P, Afzal Z. Ibuprofen and/or paracetamol (acetaminophen) for pain relief after surgical removal of lower wisdom teeth. Cochrane Database Syst Rev. 2013 Dec 12;2013(12):CD004624. doi: 10.1002/14651858.CD004624.pub2. PMID 24338830
- [Background] Bailey E, Kashbour W, Shah N, Worthington HV, Renton TF, Coulthard P. Surgical techniques for the removal of mandibular wisdom teeth. Cochrane Database Syst Rev. 2020 Jul 26;7(7):CD004345. doi: 10.1002/14651858.CD004345.pub3. PMID 32712962

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-04-30): https://cdn.clinicaltrials.gov/large-docs/34/NCT06823934/Prot_SAP_000.pdf